CLINICAL TRIAL: NCT05336981
Title: Effect of Photobiomodulation for Patients With Xerostomia
Acronym: xeros
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pia Lopez Jornet (Other)
Responsible Party: Sponsor-Investigator, Pia Lopez Jornet, Head Oral Medicine, Universidad de Murcia
Organization: Universidad de Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University Murcia 1229/2015
Record Dates: First submitted 2022-04-05; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Photobiomodulation; Low-Level Light Therapy
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Level Light Therapy ACTIVE (Experimental): Patients will receive applications of photobiomodulation directly in the region extraoral of the salivary glands ( parotid and submaxilar) will be given once a week for another 6 weeks.
  Interventions: Radiation: Low-Level Light Therapy
- Low-Level Light Therapy sham (Sham Comparator): Patients will receive applications of photobiomodulation sham directly in the region extraoral of the salivary glands ( parotid and submaxilar) will be given once a week for another 6 weeks
  Interventions: Radiation: Low-Level Light Therapy

INTERVENTIONS:
Radiation: Low-Level Light Therapy — The method consists of the application extraoral of low-intensity infrared laser in the major salivary glands-parotid, submandibular

SUMMARY:
Hyposalivation is a condition represented by a reduced salivary flow and may include symptoms such as mouth dryness (xerostomia), pain, loss of taste,dysphagia, and dysphonia, all of which greatly affect an individual's quality of life.

The aim of the present study was analized the effects of low-level light therapy irradiation (photobiomodulation PBM) on salivary gland function in patients with hyposalivation

DETAILED DESCRIPTION:
Inclusion criteria -the inclusion criteria for participating in the study were: age over 18 years; continuous xerostomia for over three months; and/or altered sialometry findings at baseline (salivary flow < 0.1 mL/min).

Exclusion criteria. : xerostomia as secondary to radiotherapy; patients with decompensated systemic disorders or cognitive problems

The 60 individuals will be randomized in 2 groups: Group A (30 individuals submitted to treatment with a PBM) and Group B (30 individuals submitted to simulated PBM). A total of 60 patients with xerostomia were enrolled in the study and cited once a week for a period of 6 weeks treatment with diode laser (810nm, 6J/cm2) or sham treatment (according to the group).

ELIGIBILITY:
Inclusion Criteria:

* the inclusion criteria for participating in the study were: age over 18 years; continuous xerostomia for over three months; and/or altered sialometry findings at baseline (salivary flow < 0.1 mL/min).

Exclusion Criteria:

* The exclusion criteria were: xerostomia as secondary to radiotherapy; patients with decompensated systemic disorders or cognitive problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
xerostomia | Change (in centimeters measured on a Visual Analogue Scale) determined between day 0 and day 15 and 45 days
  Comparison of changes in mouth Dryness Score
SIALOMETRY | before and after 45 days the procedure of laser therapy
  Sialometry was performed using the passive droll technique.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Lopez Jornet, Principal Investigator — Universidad de Murcia
Locations (2):
- Spain (2):
  - Lopez-Jornet Pia, Murcia, N/A = Not Applicable
  - Pia Lopez Jornet, Murcia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalhori KAM, Vahdatinia F, Jamalpour MR, Vescovi P, Fornaini C, Merigo E, Fekrazad R. Photobiomodulation in Oral Medicine. Photobiomodul Photomed Laser Surg. 2019 Dec;37(12):837-861. doi: 10.1089/photob.2019.4706. PMID 31873066
- [Background] Brzak BL, Cigic L, Baricevic M, Sabol I, Mravak-Stipetic M, Risovic D. Different Protocols of Photobiomodulation Therapy of Hyposalivation. Photomed Laser Surg. 2018 Feb;36(2):78-82. doi: 10.1089/pho.2017.4325. Epub 2017 Oct 12. PMID 29022754